CLINICAL TRIAL: NCT02246387
Title: Does the Manchester Operation for Pelvic Organ Prolapse Give Sufficient Apical Fixation?
Brief Title: Follow-up Study After Manchester Operation for Pelvic Organ Prolapse
Acronym: MAP-POP
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Sissel Oversand, MD, Oslo University Hospital
Other Study IDs: 2013/2093/REK
Record Dates: First submitted 2014-09-11; First posted 2014-09-22 (Estimated); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Pelvic Organ Prolapse
Keywords: Pelvic Organ Prolapse; Gynecologic Surgery Procedures; Treatment Outcome
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Manchester Operation: Manchester Operation: Native tissue repair
  Interventions: Procedure: Manchester Operation

INTERVENTIONS:
Procedure: Manchester Operation — A 3- compartment native tissue repair procedure for Pelvic Organ Prolapse.

SUMMARY:
Native tissue repair for pelvic organ prolapse (POP) is the predominant surgical technique in the investigators department and the Manchester operation the preferred procedure. The investigators long-term reoperation rates for pevic organ prolapse are very low, as documented in the investigators previous long-term follow-up study (Oversand et al, International Urogynecology Journal 2013), however the data were retrospective and patients with avulsions of the levator ani muscle were not identified. The investigators hypothesize that correct fixation and elevation of the vaginal apex, as part of a three-compartment repair procedure, is essential in the POP surgical repair, also when treating women with levator ani avulsions.

The purpose of this study is to:

* prospectively evaluate if cardinal/sacrouterine ligament plication (as part of the 3-compartment Manchester procedure) gives an adequate elevation and fixation of the vaginal apex.
* assess changes in subjective symptoms between the preoperative evaluation and the 1 and 5-year postoperative evaluations.
* evaluate whether the patients identified with levator avulsions in the investigators population have an increased risk of failure (objectively and subjectively).

DETAILED DESCRIPTION:
Many studies have shown high recurrence rates after POP surgical repair using native tissue techniques, and this led to the introduction of synthetic meshes in vaginal repair in the early 2000s. However the use of mesh has recently been put under scrutiny due to a high risk of complications, such as mesh exposure. The gran majority of the investigators patients are operated with native tissue repairs, about 60% of them by a Manchester procedure, where ligament plication is an essential part of the procedure. The investigators previous study documented high patient satisfaction and low risk of recurrence, but the data available were mainly collected retrospectively and no data were available on possible levator avulsions. Lateral defects caused by avulsions of the levator ani muscle represent a special sub-group amongst patients with POP, and are shown in several studies to have higher recurrence rates. There is no consensus on how to best repair a lateral defect in a POP, but since the prevalence of levator avulsions in patients with POP is shown to be high, the investigators find it credible that the Manchester Operation can give good results .

The main justification for this study is that the investigators already have identified a surgical technique that has documented excellent results, but studies with more detailed data quality are needed in order to better evaluate the procedure's advantages and potential disadvantages. As the use of mesh in vaginal surgery has shown unacceptable high risks of new and serious complications, there is an international focus and interest in traditional native tissue repairs and how to optimize their performance.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥ 18 years, understanding and reading Scandinavian or English language and being able to sign an informed consent. Non- Scandinavian speakers can be enrolled in the study as long as they understand and can communicate in English or Norwegian.
* Subjective distress from pelvic organ prolapse
* Cystocele Stage I - III with descent of the cervix Stage I-III, with or without a defect of the posterior wall (rectocele, enterocele, hypotrophic perineum).

Exclusion Criteria:

* Previous total hysterectomy (including removal of the cervix and the cardinal ligaments) or previous subtotal hysterectomy (removal of copus uteri).
* Previous surgery for POP
* Patients with a true Uterine prolapse with a descent of the corpus uteri stage II-III and not just an elongated cervix, as this group may benefit from other procedures than a Manchester operation (vaginal hysterectomy and sacrospinous fixation)
* Unable to understand patient information (in Norwegian or English) and sign an informed consent.
* Patients in whom a colpocleisis (closing of the vagina) is deemed the better surgical treatment, such as in elderly women not sexually active and not interested in future vaginal intercourse.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Women referred to out outpatient clinic for surgery for pelvic organ prolapse.
Sampling Method: Non-Probability Sample
Enrollment: 209 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2018-01 (Actual); Study Completion 2023-01 (Actual)

PRIMARY OUTCOMES:
Percentage with POP-Q point C equal to or less than -5 at the 1 and 5 year postoperative control compared to preoperative findings for the whole population vs subgroup with levator avulsions. | Up to 7 years
Changes in point C and D at the 1 and 5 year postoperative control compared to preoperative findings for the whole population vs subgroup with levator avulsions. | Up to 7 years

SECONDARY OUTCOMES:
Subjective satisfaction at the 1 and 5 year postoperative control (whole population vs subgroup with levator avulsions). | Up to 7 years
Changes in dyspareunia between the preoperative evaluation and at the 1 and 5 year postoperative control (whole population vs subgroup with levator avulsions). | Up to 7 years
De novo urinary incontinence at the 1 and 5 year postoperative control (whole population vs subgroup with levator avulsions). | Up to 7 years

CONTACTS AND LOCATIONS:
Overall Officials: Sissel H Oversand, MD, Principal Investigator — Oslo University Hospital; Anne C Staff, PhD, Study Chair — Oslo University Hospital; University of Oslo; Rune Svenningsen, PhD, Study Director — Oslo University Hospital; University of Oslo
Locations (1):
- Gynekologisk avdeling, Oslo Universitetssykehus Ullevål, Oslo, Norway